CLINICAL TRIAL: NCT03943329
Title: Trial of a Distal Targeting System for Cephalomedullary Nails as Part of Surgical Repair of Hip and Femoral Shaft Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-01951
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Hip Fractures; Femoral Shaft Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Procedure: Standard of Care
- Distal Targeting Treatment (Experimental)
  Interventions: Procedure: Distal targeting device technique of distal screw placement

INTERVENTIONS:
Procedure: Standard of Care — Will receive the standard of care "free-hand" technique of distal screw placement, as treated by Dr. Egol or Dr. Tejwani.
  Arms: Standard of Care
Procedure: Distal targeting device technique of distal screw placement — The second group will be the interventional group which will use the distal targeting device technique of distal screw placement and will be treated by Dr. Konda and Dr. Leucht. All relevant data to the study will be collected intra-operatively.
  Arms: Distal Targeting Treatment

SUMMARY:
This study will be a prospective, case - control trial looking at the use of a previously FDA approved device made by Stryker, a distal targeting system that eases the distal targeting of screws in cephalomedullary nails in hip and femoral shaft fractures. Patients who consent to participate in the study will either be in the control or device arm of the study depending on their surgeon.

DETAILED DESCRIPTION:
Surgeries conducted by Dr. Konda or Dr. Leucht will be done using the device technique, surgeries completed by Dr. Egol or Dr. Tejwani will be done without the device, "free hand" technique. Each arm of the study will contain 29 patients. Patients who consent to participation will be enrolled in the study and placed in the correct arm based on who their surgeon is. Demographic and injury data will be collected. Intra-operatively, control patients will receive the SOC procedure. Device arm patients will have the distal targeting device used in their procedure, but the implant, will not be different than SOC.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be greater than or equal to 18 years of age.
* The patient must have sustained a hip or femur fracture that is indicated for cephalomedullary nailing as the primary and definitive treatment measure.
* The patient must be medically cleared for operative fixation of their fracture.

Exclusion Criteria:

* The patient does not meet all of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Change in mean intra-operative radiation exposure to patients during their cephalomedullary nailing procedure. | Baseline, 1 Day

SECONDARY OUTCOMES:
Change in mean length of time to distal screw placement | Baseline, 1 Day
Change in total operative time | Baseline, 1 Day
Change in total operative cost ($) | Baseline, 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit Konda, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States